CLINICAL TRIAL: NCT03165240
Title: Randomised, Double-blind, Placebo-controlled (Within Dose Groups) and Active Controlled (Eplerenone Group) Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 3 Oral Doses of BI 690517 Over 28 Days in Female and Male Patients With Diabetic Nephropathy
Brief Title: This International Study Tests BI 690517 in Patients With Diabetic Kidney Disease. The Study Tests How 3 Different Doses of BI 690517 Are Taken up in the Body and How Well They Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1378-0008; 2017-000563-32 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- BI 690517 Dose 1 (Experimental)
  Interventions: Drug: BI 690517
- BI 690517 Dose 2 (Experimental)
  Interventions: Drug: BI 690517
- BI 690517 Dose 3 (Experimental)
  Interventions: Drug: BI 690517
- Eplerenone (Experimental)
  Interventions: Drug: Eplerenone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 690517 — Film-coated tablet
  Other Names: Vicadrostat
  Arms: BI 690517 Dose 1; BI 690517 Dose 2; BI 690517 Dose 3
Drug: Eplerenone — Film-coated tablet
  Arms: Eplerenone
Drug: Placebo — Film-coated tablet
  Arms: Placebo

SUMMARY:
The primary objective of this current trial is to investigate the safety and tolerability of 3 oral doses of BI 690517 over 28 days in female and male patients with diabetic nephropathy as add-on-therapy to Angiotensin Converting Enzyme inhibitor [ACEi] or Angiotensin-receptor blockers [ARB].

Secondary objective is to evaluate the change from baseline in Urine Albumin-to-Creatinine Ratio [UACR].

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Male or postmenopausal (last menstruation ≥ 2 years ago) patients, or female patients who are sterilized by either hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy. Male patients with partners of child-bearing potential must be willing to use condoms from the time of the first intake of study drug until follow-up.
* eGFR (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) ≥ 20 and < 75 ml/min/1.73 m2 at Visit 1 measured by the central laboratory and no planned start of renal replacement therapy during the trial.
* UACR ≥ 200 and <3500 mg/g in spot urine (midstream urine sample) at Visit 1 measured by the central laboratory.
* Treatment with either ACEi or ARB, stable dose since ≥ 4 weeks before Visit 1 with no planned change of the therapy.
* Patients with type 1 or type 2 diabetes mellitus, diagnosed before informed consent and treated with insulin, glucagon-like peptide (GLP) 1 agonists and/or oral antidiabetic medication. Treatment should have been unchanged (investigator's judgment) within 4 weeks before Visit 1 and until randomisation.
* Glycated Haemoglobin (HbA1c) < 10.0% at Visit 1 measured by the central laboratory.
* Seated SBP ≥ 110 and ≤ 180 mmHg and DBP ≥ 70 and ≤ 110 mmHg at Visit 1
* Age at screening ≥ 18 years for male and permanently sterilized female patients and ≥ 45 years for postmenopausal female patients.
* Body Mass Index (BMI) ≥ 18.5 and < 45 kg/m2.

Exclusion Criteria:

* Treatment with with SGLT2 inhibitors and/or inhibitors of aldosterone mediated effects like mineralocorticoid receptor antagonists at visit 1 and thereafter.
* Intake of potassium sparing diuretics like amiloride or potassium supplements during the study (this period starts at Visit 1).
* At Visit 1 cortisol peak level 30 minutes (± 5 min) after iv injection of Adrenocorticotropic hormone (ACTH) is an increase by less than 200 nmol/l compared to pre-ACTH injection.
* Dual or triple blockade of the Renin Angiotensin System (RAS) (e.g. ACEi + ARB; ACEi + renin inhibitor; or ARB + renin inhibitor; or ACEi + ARB + renin inhibitor) 12 weeks before Visit 1 and for the duration of study.
* History of non-diabetic renal disease according to investigator's opinion and/or renal transplant recipients.
* Hyperkalaemia (K+ > 5.0 mmol/L) at visit 1 and until start of treatment measured by any local or central lab.
* Clinical signs of acute or chronic urinary tract infection 14 days before randomization (based on investigator's judgement).
* Acute febrile diseases 14 days before randomisation (based on investigator´s judgement).
* Heart failure, patients with NYHA III / IV.
* Surgery or trauma with significant blood loss or blood donation within 12 weeks prior to first administration of study medication (based on investigator´s judgement) or planned surgeries during the trial e.g. hip replacement (based on investigator's judgement).
* Any other medical condition that in the investigator's opinion poses a safety risk for the patient or may interfere with the study objectives.
* Any laboratory value more than 3 times above upper limit normal (ULN) at screening (visit 1) or any other laboratory value outside the reference range and clinically relevant in the investigator's judgment.
* Medical history of cancer or treatment for cancer in the last two years prior to Visit 1 (except appropriately treated basal cell carcinoma of the skin, in situ carcinoma of uterine cervix, and prostatic cancer of low grade [T1 or T2] is exempted).
* Previous enrolment in this trial.
* Currently enrolled in another investigational device or drug study, or less than 30 days since ending another investigational device or drug study(s), or receiving other investigational treatment(s).
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable study patient or unlikely to complete the trial.
* Women of childbearing potential
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with drug related Adverse Events (AEs) | Up to 35 days

SECONDARY OUTCOMES:
Change from baseline in log transformed Urine Albumin-to-Creatinine Ratio (UACR) measured in morning void urine | Up to 28 days
Change from baseline in log transformed Urine Albumin-to-Creatinine Ratio (UACR) measured in daytime (10-hour) urine | Up to 28 days

CONTACTS AND LOCATIONS:
Locations (40):
- Denmark (4):
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Kolding Sygehus, Kolding
  - Bispebjerg og Frederiksberg Hospital, København NV
  - Copenhagen University Hospital, Rigshospitalet, København Ø
- France (5):
  - HOP d'Angers, Angers
  - HOP Michallon, La Tronche
  - HOP Bichat, Paris
  - HOP la Milétrie, Poitiers
  - HOP Nord Laënnec, Saint-Herblain
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - InnoDiab Forschung GmbH, Essen
  - Inamed GmbH, Gauting
  - Medizinische Hochschule Hannover, Hanover
  - Profil Institut für Stoffwechselforschung GmbH, Neuss
- Greece (4):
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - Iatriko of Athens Group/ Iatriko of P. Faliro, P. Faliro
  - Iatriko Psychikou, Psychikó
  - University General Hospital of Thessaloniki AHEPA, Thessaloniki
- Portugal (5):
  - Hospital Dr. Nélio Mendonça, Funchal
  - APDP - Associação Protectora dos Diabéticos de Portugal, Lisbon
  - CHULN, EPE - Hospital de Santa Maria, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Centro Hospitalar Universitário do Porto, EPE - Hospital de Santo António, Porto
- Russia (4):
  - Res.Inst.-Compl.Iss.Cardi.Dis., Kemerovo
  - City Clinical Hospital named after V.P. Demikhova Department of Health of Moscow, Moscow
  - Nonstate Private Healthcare Institution "Scientific Clinical Center of LLC Russian Railways", Moscow
  - Baltic Med,LLC Clinic BaltMed Ozerki, Saint Petersburg
- D & R s.r.o., Košice, Slovakia
- Spain (7):
  - Hospital A Coruña, A Coruña
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Puerta de Hierro, Majadahonda
  - Hospital Virgen Macarena, Seville
  - Hospital Clínico de Valencia, Valencia
- Sweden (4):
  - CTC Sahlgrenska Universitetssjukhuset, Gothenburg
  - Sjukhuset, Härnösand, Härnösand
  - Universitetssjukhuset, Örebro, Örebro
  - CTC Clinical Trial Consultants AB, Uppsala
- University Hospital of Wales, Cardiff, United Kingdom